CLINICAL TRIAL: NCT00857376
Title: Dose Ranging Study of the Effects of Alpha Lipoic Acid on Oxidative Stress
Acronym: Alpha
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Jarrow Formulas Inc (Industry)
Responsible Party: Principal Investigator, Pamela Ouyang, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: NA00016646; Grant # 1R21 AT003862-01A2
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome
Keywords: Heart disease risk factors; Risk factor management; Pre-Diabetes; Hypertension; obesity; glucose intolerance; high cholesterol; abdominal obesity; enlarged waist
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Hypertension; Obesity; Hypercholesterolemia; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): Placebo 2 tabs three times daily
  Interventions: Dietary Supplement: Alpha lipoic acid at 3 doses compared to placebo
- Alpha lipoic acid 1 (Experimental): Alpha lipoic acid 600 mg daily
  Interventions: Dietary Supplement: Alpha lipoic acid at 3 doses compared to placebo
- Alpha lipoic acid 2 (Experimental): Alpha Lipoic acid 1200 mg daily
  Interventions: Dietary Supplement: Alpha lipoic acid at 3 doses compared to placebo
- Alpha lipoic acid 3 (Experimental): Alpha lipoic acid 1800 mg daily
  Interventions: Dietary Supplement: Alpha lipoic acid at 3 doses compared to placebo

INTERVENTIONS:
Dietary Supplement: Alpha lipoic acid at 3 doses compared to placebo — This is a randomized study comparing the antioxidant effects of 3 doses of alpha lipoic acid (total of 600 mg daily, 1200 mg daily and 1800 mg daily) compared to placebo. These doses will be taken as 2 pills 3 times a day for 8 to 10 weeks.

SUMMARY:
Heart disease is the most common cause of death in the United States and it is commonly found in people with diabetes and high cholesterol. Inflammation is one mechanism by which diabetes and elevated cholesterol damage blood vessels. Inflammation can be increased by oxidative stress. This study will see if Alpha Lipoic acid, a potent antioxidant and over the counter product, reduces blood levels of markers of oxidative stress and inflammation when compared with placebo. Placebo is a substance that looks like the real product, but contains no active product.

DETAILED DESCRIPTION:
This is a randomized study. A randomized study means you will be assigned by chance (like the toss of a coin) to one of four groups and receive either alpha lipoic acid (ALA or placebo (an inactive substance that looks like the real drug). In this study, there is a 1 out of 4 chance you will receive placebo. Three of the groups will receive different doses of ALA and one group will receive placebo only. The groups are: placebo only, 600 mg ALA, 1200 mg ALA, and 1800 mg ALA a day. At some point all study participants will receive placebo; sometimes the pills will be ALA and sometimes they will be placebo. You will not know which you are taking on any given day.

This study is also double-blinded, which means that you, the study doctor, and the Sponsor will not know until the end of the study whether you are receiving ALA or placebo only. Your study doctor can find out if you are receiving ALA or placebo if needed in an emergency.

If you agree to be in this study, you will be asked to come in for up to 6 visits in 12 weeks. You should be fasting before some of these visits. Fasting means that you should have nothing to eat or drink, except water with your usual morning medications, for 10 hours before your scheduled study visit. The study staff will go over this with you each time.

Visit 1-Screening: (about 3 hours)

• Please fast before this visit

In order to find out if you qualify to take part in the study, you will have the following tests and procedures done during this visit including:

* Your health history will be taken
* Your height, weight, and blood pressure will be measured
* You will have an electrocardiogram (ECG)
* You will give fasting blood samples of about 3-5 tablespoons and urine samples
* If you are female and can have children, you will be given a urine pregnancy test
* You will take a glucose tolerance test (GTT) A dietitian will briefly discuss your diet and exercise. An ECG will be done to measure your heart function. ECG measures the electrical activity of your heart. You will be asked to lie down and small sticky pads will be placed on your arms, legs, and across your chest.

The GTT test involves collecting 1 blood sample before, and 4 samples up to 2 hours after, you drink a measured amount of glucose (a sugar) in a pleasant tasting liquid. You will have 2 tablespoons of blood drawn. An indwelling intravenous (IV) needle will be inserted into your vein for the 2-hour period so that individual needle sticks will not be needed.

Depending on the results of your blood and urine tests, you may be asked to come in for a second visit in about 1 week. The screening blood tests may provide you with information on your health that could be important to you, for example diagnosing diabetes.

VISIT 2: (about 1 hour)

• You do not have to fast for this visit and may take your morning medications as usual

You will have the following tests and procedures done during this visit including:

- You will meet with a dietician for an assessment of your eating habits. The dietitian will advise you on how to maintain a stable diet during the study.

* If your blood tests indicate that you have diabetes, you will receive instructions on diet and exercise to improve your blood sugar levels.
* If your HbA1c level is high, you will be given a home glucose monitoring device (glucometer) with instructions on its use for daily testing. HbA1c is a measure of average glucose levels over the prior few weeks.
* You will be given a 2-week supply of study drug and asked to stop any over- the-counter vitamins that you are taking until you have completed this study. We will provide 3 bottles of study medicine at a time. Each bottle will be uniquely identified for use in the morning, midday or evening. You will be asked to take 2 tablets from the morning bottle, then 2 from the midday bottle and 2 from the evening bottle. You will also be given a daily multivitamin to take. This will be a total of 7 tablets a day for 10 weeks.

All unused study drug should be returned when you come in for the next visit in 2 weeks. It is important that you are able to take all the study drug. If we find that you are unable to take most of the study drug, you will be removed from the study.

VISIT 3: (about 6-8 hours)

•

* Please be fasting and do not have alcohol or exercise for 48 hours prior to the visit. You may be asked to withhold some of your usual medicines on this day but bring the doses to the visit with you to be taken at a later time. You will have the following tests and procedures done during this visit including:
* Brachial artery ultrasound: This is a way to see how the walls of your arteries respond to change in blood flow. For this test, you will lie on a bed and we will take sound wave pictures of the artery in your elbow area. After the initial pictures, we will then inflate a blood pressure cuff on your upper arm for 5 minutes. As soon as the cuff is deflated more pictures of the same artery are taken. We will give then give you a pill called nitroglycerine to dissolve under your tongue. When the pill dissolves in a few minutes, final pictures of the same artery will be taken.
* The brachial test will be repeated 2 hours after a high fat meal is eaten. We will give the meal to you It will contain known amounts of fat,carbohydrates, and protein.
* Augmentation index: This is a test to see how stiff the walls of your artery may be. A small microphone will record the signal from the artery in your wrist for about 5 minutes.
* Several samples of blood (2 tablespoons) will be taken before you eat the high fat meal and when the second brachial test is completed. An indwelling IV needle may be inserted into your vein during this period so that individual needle sticks will not be needed.
* DEXA scan. DEXA is a 4-5 minute x-ray body scan that provides accurate body fat mass measurements.If you are a woman who can have children, you will have a urine pregnancy test. If you are pregnant you will NOT be able to have the DEXA scan.
* A dietician will assist you with food questionnaire about your usual diet.
* A 4-week supply of study drug will be given to you with instructions on how to take it. Please bring any remaining study drug bottles with you to your next visit.

Visit 4: telephone call. You will also be asked about your ability and willingness to continue to take the study medicine until the end of the study.

We will also ask if you are having any new symptoms that may indicate low blood sugar such as hunger, shakiness, dizziness, confusion, difficulty speaking, feeling anxious or weak.

You should notify the study team at any time by telephone to report these symptoms. You may be asked to come in for an extra visit if these are occurring.

Visits 5(day 1 and 2 final visits): (about 4 hours each day for 2 days)

• Please be fasting and do not have alcohol or exercise for 48 hours prior to these visits. You may be asked to withhold some of your usual medicines on both days but bring the doses to the visit with you to take at a later time.

These 2 visits may be done on 2 consecutive mornings.

Visit 5 day 1

You will have a brachial artery ultrasound with nitroglycerine, a DEXA scan, a 2 hour GTT blood test with an indwelling IV needle in your vein, height, weight, blood pressure.

- If you are a woman who can have children, you will be given a urine pregnancy test. If you are pregnant, you will NOT be able to have the DEXA scan that is part of this visit.

Visit 5 day 2

The brachial ultrasound will be repeated after a high fat meal is eaten which is provided by the study center.

You will have blood samples taken before and after the test and you will also meet with a dietitian for a final food questionnaire.

- You will return any unused study drug bottles.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or more yrs,
* Are able to give informed consent
* Diabetic on stable doses of oral medications or diet or
* Metabolic syndrome defined as having 3 or more of the following:
* Impaired or fasting glucose > or = 100 mg/dL) or impaired glucose tolerance
* Waist circumference > 40 inches in men and > 35 inches in women,
* Hypertension (> or = 130/85 mmHg) or are on antihypertensive medication,
* LDL < or = 50 mg/dL in females and < or = 40 mg/dL in men,
* Triglyceride > or = 150 mg/dL

Exclusion Criteria:

* Are on oral hypoglycemic drugs or insulin with HbA1c > 7.5,if diabetic,
* On antioxidant supplementation and are unable or unwilling to stop,
* A woman on hormone replacement therapy,
* On medications that may have antioxidant or anti-inflammatory effects or effects on insulin sensitivity, e.g. HMGCo-A reductase inhibitor that cannot be discontinued for the duration of the study,
* Current smoker (within 3 months prior to enrollment),
* Have known coronary artery disease or stroke,
* Have other diseases associated with active inflammation e.g. connective tissue disease, malignancy,
* have a CRP > or = 10 mg/dl on screening blood with clinical evidence of inflammation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
This study will provide information on the effect of a dose range of ALA on oxidative stress biomarkers. | 3 months

SECONDARY OUTCOMES:
To determine whether ALA improves vascular function through its effects on oxidative stress | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ouyang, MBBS, Principal Investigator — Johns Hopkins University